CLINICAL TRIAL: NCT05853627
Title: Mismatch vs. Standard Intervention During Memory Reconsolidation Blockade With Propranolol: Effect on Psychophysiological Reactivity During Traumatic Imagery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kaloyan Tanev, MD, Senior Director of Research, The Home Base Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1R21MH131987-01A1 (NIH)
Record Dates: First submitted 2023-04-20; First posted 2023-05-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: The efficacy of the MM intervention will be contrasted with a standard (STD) reactivation condition that does not include an intentional MM component. We will randomize ndividuals who have experienced a traumatic event and meet our entry criteria (please see research strategy) to one of the two treatment arms: STD/PPNL and MM/PPNL. Participants' psychophysiological (heart rate, skin conductance, corrugator electromyogram (EMG)) responses during script driven imagery of their traumatic event will constitute the R21 target.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned to the STD vs. MM condition. The psychophysiology assessor, who will perform the data analysis, will be blind to Condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mismatch reactivation condition (Experimental): The participant will recite their trauma narrative to the psychologist for 10-20 minutes. However, during each recitation, a "mismatch" condition, different for each session, will be added to the reactivation procedure by having the participant do the following (in order of sessions.
  Interventions: Behavioral: Memory reactivation procedures; Drug: Propranolol
- Standard reactivation condition (Active Comparator): The intervention will be the same for each of the six intervention sessions. The participant will recite to the psychologist the narrative they previously composed for 10-20 min. The psychologist will congratulate the participant for having succeeded in this task and advise them they are finished for the day.
  Interventions: Behavioral: Memory reactivation procedures; Drug: Propranolol

INTERVENTIONS:
Behavioral: Memory reactivation procedures — In the Mismatch condition, a different, unexpected mismatch will be incorporated into the reactivation. In the Standard condition, the participant will read the narrative the same way each time.
Drug: Propranolol — Propranolol will be administered 60-min prior to each of six weekly 10-20 min. traumatic memory reactivation sessions.

SUMMARY:
The proposed R21 project will attempt to further develop a novel intervention for posttraumatic stress symptoms inspired by the science of memory reconsolidation. Work in normal humans has shown that when a stable, consolidated memory is reactivated (i.e., retrieved) under appropriate conditions, it reverts to an unstable state, a process referred to herein as deconsolidation. In such a state, the memory is susceptible to the action of various "amnestic" agents that may inhibit its reconsolidation, thereby weakening it. The β-adrenergic blocker propranolol (PPNL) possesses such amnestic properties. More recent research has found that in order to initiate deconsolidation, there must be a prediction error, or mismatch, between what is expected and what occurs when the memory is reactivated.

Prior placebo-controlled, randomized clinical trials (PBO-RCT) from our laboratory have found that when propranolol is administered concomitant with the reactivation of a psychologically traumatic memory, the memory is weakened, as revealed by subsequent lower physiological (heart rate, skin conductance, facial electromyogram) responding during script-driven mental imagery. Clinical applicability was evaluated in a PBO-RCT, in which PTSD participants receiving propranolol underwent six weekly sessions of 10-20 min of "standard" (STD) traumatic memory reactivation stimulated by reading a narrative. At post-treatment, these participants showed a greater reduction of PTSD symptoms compared to participants who had taken PBO. The goal of the proposed study is to test whether intentionally incorporating innovative mismatch (MM) into traumatic memory reactivation can improve upon physiological responding during script-driven mental imagery.

Participants will be randomized to one of 2 treatment arms: STD/PPNL and MM/PPNL. A baseline assessment will measure psychophysiological responsivity to script-driven mental imagery (target measure). PPNL will be administered 90-min prior to each of six weekly 10-20 min. traumatic memory reactivation sessions. In the MM condition, a different, unexpected mismatch (e.g., singing the narrative) will be incorporated into the reactivation. In the STD condition, the participant will read the narrative the same way each time. The focus of the R21 proposal will be to assess whether the MM/PPNL group shows lower subsequent physiological responses than the STD/PPNL group

DETAILED DESCRIPTION:
The proposed project under the R21 Basic Experimental Studies Involving Humans (BESH) mechanism aims to test whether adding 'mismatch' (MM) to traumatic memory reactivation under the influence of the beta-(nor)adrenergic blocker propranolol (PPNL), compared to no mismatch reactivation, further reduces physiological reactivity during script driven imagery of the traumatic event. We propose that the mechanism for the propranolol MM treatment is a) deconsolidation of the traumatic memory instigated by MM, followed by b) blockade of the reconsolidation of the memory by the amnestic agent PPNL. The efficacy of the MM intervention will be contrasted with a standard (STD) reactivation condition that does not include an intentional MM component. We will randomize individuals who have experienced a traumatic event and meet our entry criteria (please see research strategy) to one of the two treatment arms: STD/PPNL and MM/PPNL. Participants' psychophysiological (heart rate, skin conductance, corrugator electromyogram (EMG)) responses during script driven imagery of their traumatic event will constitute the R21 target.

On the initial assessment day, participant candidates will be screened for eligibility based upon the inclusion/exclusion criteria. After the candidate provides written informed consent, a doctoral-level clinician will administer the psychometric instruments. Participant candidates will complete a narrative describing the traumatic event that caused PTSD.

Based on the narrative, the psychologist will then prepare a 100-word script portraying the most salient aspect ("hot spot") of the narrative, which will be recorded for audio playback in the psychophysiology laboratory. Participants not physiologically reactive to the traumatic script will be excluded. If all of the foregoing is completed successfully, participants will be randomized to one of the two arms above.

The participant will return to the clinic one week later for the first of six weekly intervention sessions. Ninety min. prior to its commencement, the participant will ingest the study medication. The participant will then recite the narrative aloud for 10-20 min. In the STD condition, the participant will recite the narrative in an expected manner, i.e., in the same way during each session. In the MM condition, the participant will recite the narrative in an unexpected manner, different for each weekly session. Examples of unexpected conditions will include such things as reciting their narrative while skipping over each word that contains the letter "e", and reciting the narrative in a make-believe accent. A week following the final intervention session, the participant will return for the post-treatment psychophysiological testing. These will be repeated at the one-month follow-up session.

The data will be analyzed by hierarchical linear modeling and regression techniques. The projected sample sizes will provide adequate power to test the proposed study's hypotheses (see Design and Power Analysis section).

ELIGIBILITY:
Inclusion Criteria:

* Initial participants will be males or females 18-65 years old who have experienced a traumatic event that meets the DSM-5 PTSD A criterion, and whose PCL-5 score is >33 (to maximize the likelihood that they will meet our psychophysiological inclusion criterion). In order to be randomized, participants must further meet this psychophysiological inclusion criterion during baseline script-driven imagery testing Although we do not require a diagnosis of PTSD, because we have set a minimum psychophysiological inclusion criterion and a valid Criterion A traumatic event, our sample will include a substantial number, likely a majority, of PTSD participants.

Exclusion Criteria:

1. Basal sitting or standing systolic blood pressure <90/60 mm Hg or basal HR <50 BPM. Those participant-candidates excluded for this reason with such readings will be counseled and referred for further clinical consultation if symptomatic or if they wish to be referred even if asymptomatic.
2. Medical condition that contraindicates PPNL, e.g., congestive heart failure, heart block, insulin- requiring diabetes, chronic bronchitis, emphysema, or asthma. Asthma attacks will only be exclusionary if they: a) occurred within the past ten years, b) occurred at any time in life if induced by a β-blocker, or c) are currently being treated
3. Previous adverse reaction to, or non-compliance with, a β-blocker
4. Current use of medication that may involve potentially dangerous or confounding interactions with PPNL, including anti- hypertensives, antiarrhythmics, and benzodiazepines. (Possible inhibition of CYP2D6 isoenzyme-dependent reactions will not be of concern in this study, because PPNL will only be administered once a week)
5. Presence of drugs of abuse, including opiates, marijuana, cocaine, amphetamines, or alcohol at the initial assessment
6. Pregnancy or breast feeding. Women of childbearing potential will have a pregnancy test at the initial assessment
7. Presence of a contraindicating psychiatric condition, e.g., psychotic, bipolar, melancholic, or active substance use disorder; or suicidality (see below)
8. Initiation of, or change in, psychotropic medication within the previous two months. For participants receiving stable doses of pharmacotherapy, they and their clinicians-prescribers will be asked not to alter the regimen during the proposed two-month study period (excluding the one-month follow-up) except in clinically urgent circumstances. If this becomes necessary, a decision will be made on a case-by-case basis about retaining the participant or terminating participation
9. Current participation in any psychotherapy other than supportive. Participants will be asked not to initiate new psychotherapy during the proposed two-month study period (excluding the one-month follow-up) except in clinically urgent circumstances. If this becomes necessary, a decision will be made on a case-by-case basis about retaining the participant or terminating participation
10. Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation
11. Participant candidate does not understand English. This exclusion criterion is necessary because the procedures require a nuanced dialogue with English-speaking investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite score of psychophysiological reactivity (comprising heart rate, skin conductance, and electromyography of the left corrugator muscle) using the Biopac system. | Baseline (week 0)
  psychophysiological responding during script-driven traumatic imagery compared to no imagery.
Composite score of psychophysiological reactivity (comprising heart rate, skin conductance, and electromyography of the left corrugator muscle) using the Biopac system. | Post-treatment (week 7)
  psychophysiological responding during script-driven traumatic imagery compared to no imagery.
Composite score of psychophysiological reactivity (comprising heart rate, skin conductance, and electromyography of the left corrugator muscle) using the Biopac system. | Follow up (week 11)
  psychophysiological responding during script-driven traumatic imagery compared to no imagery.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Home Base Program, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No subject identifiers will be released. The results of this study will be shared with the wider scientific community. Data will be stored in the NIMH Data Archive (NDA), where it will be available for secondary analysis. Data will be findable by the research community through the NDA Collection that will be established when this application is funded. The data will be uploaded on a rolling basis and brought current twice annually following the usual NDA data submission dates. To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. For all publications, an NDA study will be created. Each of these studies will be assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication.